CLINICAL TRIAL: NCT02816931
Title: Plasma Drug Concentrations in the Treatment of Multidrug-resistant Tuberculosis in Relation to Minimum Inhibitory Concentrations - a Prospective Observational Study
Brief Title: Drug Concentrations in the Treatment of MDR-TB Related to Minimum Inhibitory Concentrations
Acronym: TDM-MDR-TB
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Fudan University (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Judith Bruchfeld, Senior Consultant, Associate Professor, Karolinska Institutet
Other Study IDs: 540-2013-8797; D0879701 (Other: Swedish Research Council)
Record Dates: First submitted 2016-04-14; First posted 2016-06-29 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Tuberculosis, Multidrug Resistant
Keywords: Treatment; Drug Monitoring; Minimum Inhibitory Concentration; Dried Blood Spot Method; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mycobacterium tuberculosis isolates will be frozen and stored for whole genome sequencing in order to compare with clinical and phenotypic characteristics. Blood samples will be frozen and stored for drug concentration analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Multi-drug resistant tuberculosis (MDR-TB) is steadily increasing world-wide, urging for the need of improved treatment strategies. In order to protect the few available drugs that are left, ensuring adequate plasma concentrations of the drugs are important. Individualized therapy using plasma drug concentrations and minimal inhibitory concentration (MIC) determination may be of importance (1). The plasma drug concentrations and the MICs of the second-line drugs will be compared, aiming at increasing the knowledge about pharmacokinetic/pharmacodynamic (PK/PD) indices in the treatment of MDR-TB. In the future, the aim is an individualised therapy, where sub-therapeutic drug concentrations can be adjusted by the use of therapeutic drug monitoring (TDM). TDM in the treatment of MDR-TB may improve clinical outcome for the patients, but plasma concentrations must be assessed together with clinical and microbiological factors (2).

In this observational study the hypothesis is that the ratio between drug concentrations and MICs of the anti-tuberculous drugs, are correlated to the time to sputum culture conversion, the bacterial load measured as time to positive liquid culture (TTP) and clinical outcome. Consenting adult patients with pulmonary MDR-TB patients in China will be recruited. MIC-determination of Mycobacterium tuberculosis will be performed in BACTEC 960 MGIT and drug concentration will be determined at 2, 4 and 8 weeks after treatment initiation using liquid chromatography tandem mass spectrometry (LC-MS/MS), simultaneously assessing Dried Blood Spot (DBS) as a bio-sampling method. Sputum cultures will be obtained regularly throughout the treatment to measure the time to culture positivity (TTP). Clinical follow up according to WHO criteria will be performed at the end of treatment completion.

DETAILED DESCRIPTION:
Consenting adult patients with active pulmonary MDR-TB in the study hospital in China (n=50), will be included in the study. Detailed demographic background information as well as baseline clinical characteristics will be collected. Sputum samples for culture and Time to culture positivity (TTP) will be collected at inclusion and at day 2, 7 and week 2, 4, 8 and 12 weeks after start of treatment. MIC-determination of Mycobacterium tuberculosis for all drugs included in the patient's treatment, will be performed mainly using Sensititre TREK kit, complemented with BACTEC 960 MGIT when necessary. After two weeks of TB-treatment, plasma drug concentrations of all the drugs used will be collected. Multiple blood samples (0, 1, 2, 4, 6, 8 and 10 h after drug intake) will be collected in order to accurately calculate the free area under the time-versus concentration curve (fAUC) and maximum concentrations (fCmax). The exposure variables are the fAUC and the fCmax and their ratio with the MIC for the bacteria of the different drugs. Furthermore, blood sampling to assess stability of drug concentrations will be performed at week 8 and week 12 (0, 4 and 6 h post-dose). In order to evaluate if low ratios of fAUC/MIC and fCmax/MIC are associated with poor clinical outcome, clinical parameters as well as sputum culture conversion, time to culture positivity (TTP), inflammatory markers and radiological imaging will be followed up during the first three months of treatment. After treatment completion, the WHO criteria for defining treatment outcome will be applied.

Furthermore, a method of simultaneous determination using LC-MS/MS of the second-line drugs used, will be developed and compared with the use of Dried Blood Spot assay (DBS). DBS has the advantage of enabling drug concentration analysis even in remote areas, since transportation of the filter papers is easy.

ELIGIBILITY:
Inclusion Criteria:

* Active pulmonary MDR-TB tuberculosis, consenting adult

Exclusion Criteria:

* HIV, pregnancy, Extensively Drug Resistant TB (XDR-TB), unwilling to participate, critically ill such as admitted to the ICU, ongoing treatment with 5 MDR TB drugs or more for more than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients newly diagnosed with pulmonary MDR-TB admitted to the study hospital in Xiamen, China is eligible for inclusion. Phenotypic DST results identifying M. tuberculosis resistant to rifampicin and isoniazid will be performed. Patient's will be informed and asked to participate in the study both orally and in writing.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Free area under the curve (fAUC) for second-line TB drugs, separate and in relation to minimum inhibitory concentration (MIC) | after 2 weeks of treatment (rich sampling)
  Descriptive data of the distribution of fAUC of MDR-TB patients, with regard to existing recommended levels
Free maximal concentration (fCmax) for second-line TB drugs, separate and in relation to minimum inhibitory concentration (MIC) | after 2 weeks of treatment (rich sampling)
  Descriptive data of the distribution of fCmax of MDR-TB patients, with regard to existing recommended levels

SECONDARY OUTCOMES:
Sputum culture conversion | 3 months of treatment
  The proportion of patient's with sputum culture conversion after 3 months of TB treatment
Sputum culture conversion | 2 months of treatment
  The proportion of patient's with sputum culture conversion after 2 months of TB treatment
Time to sputum culture positivity (TTP) | 3 months
  Changes in the TTP during the first 3 months of treatment
Change in TB score 2 during the first 3 months of treatment | 3 months
  Decrease or increase of TB score during treatment
Changes in drug resistance - WGS (whole genome sequencing) or MIC | 3 months
  Proportion of patient's with significant changes in the drug resistance, phenotypic (MIC) and genotypic (whole genome sequencing) of the TB drugs used, for patients who are still culture positive after 3 months of treatment.
Time to sputum culture conversion | 24 months
  Time (in months) from start of treatment until the first out of two consecutive negative sputum cultures, collected at least 30 days apart.
Treatment outcome | 36 months
  Treatment outcome according to the WHO, including relapse
EQ-5D Quality of life | 3months
  Descriptive analysis of EQ-5D during MDR-TB treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hu Yi, MD Ass Prof, Study Director — Fudan University, Shanghai; Sven Hoffner, Prof, Study Chair — Karolinska Institutet; Biao Xu, Prof, Study Chair — Fudan University, Shanghai; Thomas Schön, MD Ass Prof, Study Chair — Kalmar County Hospital; Rongrong Zheng, MD, Study Chair — Xiamen CDC; Lina Davies Forsman, MD, Study Chair — Karolinska Institutet, Department of Medicine, Unit of Infectious Diseases, Stockholm; Xiangyang Yao, MD, Study Chair — Xiamen First Affiliated Hospital; Jan-Willem Alffenaar, Prof PhamD, Study Chair — University Medical Center of Groningen; Remco Koster, PhamD PhD, Study Chair — University Medical Center of Groningen; Katarina Niward, MD, Study Chair — University Hospital, Linkoeping; Judith Bruchfeld, MD Ass. Prof, Principal Investigator — Karolinska Institutet, Department of Medicine, Unit of Infectious Diseases, Stockholm; Jakob Paues, MD, PhD, Study Chair — University Hospital, Linkoeping; Johanna Kuhlin, MD, MSc, Study Chair — Karolinska Institutet
Locations (1):
- Xiamen Designated TB hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsultan A, Peloquin CA. Therapeutic drug monitoring in the treatment of tuberculosis: an update. Drugs. 2014 Jun;74(8):839-54. doi: 10.1007/s40265-014-0222-8. PMID 24846578
- [Background] Chigutsa E, Pasipanodya JG, Visser ME, van Helden PD, Smith PJ, Sirgel FA, Gumbo T, McIlleron H. Impact of nonlinear interactions of pharmacokinetics and MICs on sputum bacillary kill rates as a marker of sterilizing effect in tuberculosis. Antimicrob Agents Chemother. 2015 Jan;59(1):38-45. doi: 10.1128/AAC.03931-14. Epub 2014 Oct 13. PMID 25313213
- [Background] Ghimire S, Bolhuis MS, Sturkenboom MG, Akkerman OW, de Lange WC, van der Werf TS, Alffenaar JW. Incorporating therapeutic drug monitoring into the World Health Organization hierarchy of tuberculosis diagnostics. Eur Respir J. 2016 Jun;47(6):1867-9. doi: 10.1183/13993003.00040-2016. Epub 2016 Mar 17. No abstract available. PMID 26989104
- [Background] van der Burgt EP, Sturkenboom MG, Bolhuis MS, Akkerman OW, Kosterink JG, de Lange WC, Cobelens FG, van der Werf TS, Alffenaar JW. End TB with precision treatment! Eur Respir J. 2016 Feb;47(2):680-2. doi: 10.1183/13993003.01285-2015. No abstract available. PMID 26828056
- [Derived] Davies Forsman L, Niward K, Kuhlin J, Zheng X, Zheng R, Ke R, Hong C, Werngren J, Paues J, Simonsson USH, Eliasson E, Hoffner S, Xu B, Alffenaar JW, Schon T, Hu Y, Bruchfeld J. Suboptimal moxifloxacin and levofloxacin drug exposure during treatment of patients with multidrug-resistant tuberculosis: results from a prospective study in China. Eur Respir J. 2021 Mar 11;57(3):2003463. doi: 10.1183/13993003.03463-2020. Print 2021 Mar. No abstract available. PMID 33154028
- [Derived] Davies Forsman L, Niward K, Hu Y, Zheng R, Zheng X, Ke R, Cai W, Hong C, Li Y, Gao Y, Werngren J, Paues J, Kuhlin J, Simonsson USH, Eliasson E, Alffenaar JW, Mansjo M, Hoffner S, Xu B, Schon T, Bruchfeld J. Plasma concentrations of second-line antituberculosis drugs in relation to minimum inhibitory concentrations in multidrug-resistant tuberculosis patients in China: a study protocol of a prospective observational cohort study. BMJ Open. 2018 Oct 4;8(9):e023899. doi: 10.1136/bmjopen-2018-023899. PMID 30287613